CLINICAL TRIAL: NCT05642598
Title: Pilot Study of a Smartphone-Based Vaping Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pivot Health Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer Marler, MD, VP of Clinical and Medical Affairs, Pivot Health Technologies Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-503
Record Dates: First submitted 2022-11-18; First posted 2022-12-08 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Vaping Cessation
Keywords: vaping cessation; e-cigarette cessation; digital health; mobile apps; health promotion
MeSH Terms: interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pivot for Vape (Experimental): A commercially available mobile phone app and program for vaping cessation
  Interventions: Behavioral: Pivot for Vape

INTERVENTIONS:
Behavioral: Pivot for Vape — "Pivot for Vape" vaping cessation smartphone app and program

SUMMARY:
Prospective, open label, single center clinical study enrolling up to 100 participants to evaluate the effect of the Pivot vaping cessation program.

DETAILED DESCRIPTION:
This is a prospective, open label, single center clinical study conducted with IRB approval enrolling up to 100 adult participants who report daily vaping. The study will be performed remotely on an ambulatory basis.

Participants will be asked to set up and use the "Pivot for Vape" program. The program includes an app, moderated online community, and SMS-based coaching with a tobacco treatment specialist. The study duration is 52 weeks, with the estimated active time using the program of up to 6 months and the time thereafter as follow-up. Participants will receive online questionnaires at intervals throughout the study.

Potential participants will complete an online screening form. Eligible participants will be called to confirm eligibility, discuss the study, and have their questions about the study answered. Interested eligible participants will complete the electronic informed consent form and baseline questionnaire prior to downloading the app on their smartphone.

The investigators aim to assess the performance of the "Pivot for Vape" program, with a focus on assessing use and engagement, changes in attitudes towards quitting vaping and changes in vaping behavior over the course of the 1-year study, as well as participant feedback on the set-up, design, use experience, and impact of the program.

ELIGIBILITY:
Inclusion Criteria:

* Current daily nicotine vape/e-cigarette user for at least the past 30 days
* Plans to quit vaping in the next 6 months
* Reports average VSPD ≥ 5
* Interested in working with a vape cessation coach via SMS text
* Resident of the United States
* Able to read and comprehend English
* Owns and uses a smartphone compatible with the study app (iPhone 5 and above with operating system iOS 12 and above, or, Android 7.0 and above with operating system Android 7.0 and above)
* Has daily internet access on smartphone
* Comfortable downloading and using smartphone apps
* Willing to sign the Informed Consent Form (ICF)

Exclusion Criteria:

* Using other vaping cessation apps, coaching, classes, or quit programs at entry
* Currently using cigarettes
* If previous cigarette smoker, need to have quit smoking at least 3 months ago (self-report)
* Failure to provide contact or collateral information, and/or failure to verify email address
* Participation in a previous study sponsored by Pivot Health Technologies Inc. (formerly Carrot Inc.)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Vaping cessation rate: 30-day PPA | 6 months (26 weeks)
  30-day point prevalence abstinence (PPA) is defined as a participant self-report of no vaping for the past 30 days

SECONDARY OUTCOMES:
Change in expected difficulty in staying quit | 6 months (26 weeks)
  Participant self report. Difficulty staying quit (DTQ), scale 1-10, higher values indicate greater difficulty staying quit (vape free).
Change in confidence levels toward quitting vaping (expected success in quitting) | 6 months (26 weeks)
  Participant self report. Confidence levels or expected success in quitting (STQ), scale 1-10, higher values indicate greater confidence/greater expected success in quitting.
Desire to quit vaping | 4 weeks
  Desire to quit vaping defined as a participant self-report of "yes" to "Would you like to completely stop vaping/using e-cigarettes?". Answer options include "yes" and "no".
Vaping cessation rate: 7-day PPA | 6 months (26 weeks)
  7-day point-prevalence abstinence (PPA) is defined as a participant self-report of no vaping in the past 7 days.
Self-reported continuous abstinence at 26 weeks | 6 months (26 weeks)
  Defined as a self-report of 7-day (or greater) ppa at 12 weeks, self-report of 30-day ppa at 26 weeks, and no. more than 5 vaping sessions since 12 weeks.
Self-reported continuous abstinence at 52 weeks | 1 year (52 weeks)
  Defined as a self-reported continuous abstinence at 26 weeks and self-report of 30-day ppa at 52 weeks.
Self-reported serial abstinence | 1 year (52 weeks)
  Defined as a self-report of continuous abstinence at 26 weeks, a self-report of 30-day ppa at 52 weeks, and no more than 5 vaping sessions since 26 weeks.
Self-reported abstinence from all tobacco products | 6 months (26 weeks)
  Tobacco product use is self-reported. Participants are asked about the following products: cigars, cigarillos, little filtered cigars, a regular pipe, cigarettes, hookah or water pipe, smokeless tobacco, chew, and snuff
The proportion of participants who reduced their vaping sessions per day (VSPD) by ≥ 50% compared to baseline | 6, 12, 26, and 52 weeks
  Number of vape session per day (VSPD) are self-reported
Percent change in vape sessions per day (VSPD) compared to baseline | 6 months (26 weeks)
  Number of vape session per day (VSPD) are self-reported
The proportion of participants who reduced the amount of vape juice / e-liquid consumed by ≥ 50% compared to baseline | 6, 12, 26, and 52 weeks
  Vape juice / e-liquid consumption volume is self-reported in mL/day or mL/week
Percent change in the amount of vape juice / e-liquid consumed compared to baseline | 6 months (26 weeks)
  Vape juice / e-liquid consumption volume is self-reported in mL/day or mL/week
The proportion of participants who reduced their vape juice / e-liquid nicotine concentration by ≥ 50% compared to baseline | 6, 12, 26, and 52 weeks
  Nicotine concentration is self-reported in mg/mL
The proportion of participants who report decreased/unchanged/increased vaping compared to baseline | 6, 12, 26, and 52 weeks
  Amount of vaping is quantified as volume/day (mL/day) x concentration of nicotine (mg/mL)
Number of quit attempts | 4, 12, 26, and 52 weeks
  Defined as participant answering ≥1 to the following question: "Since you began the study, how many times have you tried to quit vaping where you've gone at least 1 day without vaping, even a single puff?"
Change in vaping / e-cig dependence | 12, 26, and 52 weeks
  Assessed via the Penn State Electronic Cigarette Dependence Index, 10 items. Possible scores on the index range from 0-20. Scores from 0-3 indicate no dependence, 4-8 low dependence, 9-12 medium dependence, 13+ high dependence
User feedback - starting the vaping cessation program | 2 weeks
  Specifically regarding set-up and getting started with the program. Participants asked: "How easy or difficult was it to set-up and get started in the Pivot program?". Answered on a range from 1-10; 1 = Very difficult, and 10 = Very easy. A higher score indicates greater ease of program set-up and getting started.
User satisfaction - Net Promoter Score | 4, 12, and 26 weeks
  Specifically regarding likelihood to recommend to a friend, Net Promoter Score (NPS). Participants asked: "How likely are you to recommend your study program to a friend or colleague?". Answered on a range from 1-10; 1 = Not at all likely, and 10 = Very likely. A higher score indicates greater user satisfaction and promotion of the program.
User satisfaction - helpful for quitting | 8 and 12 weeks
  Specifically regarding whether the program was useful in helping participants quit vaping. Participants are asked: "Which of the following best describes the Pivot program's ability to help someone quit vaping?". Answer choices include the following: "The program is extremely helpful to quitting vaping"; "The program is helpful to quitting vaping"; "The program does not affect being able to quit vaping"; and "The program makes quitting vaping harder".
Engagement with program - app openings | 6 months (26 weeks)
  Collected via back-end app data collection. Engagement is specifically assessed with number of times the Pivot app was opened (number of app openings), number of days the app was opened, and the number of weeks the app was opened.
Engagement with program - number of days with app openings | 6 months (26 weeks)
  Collected via back-end app data collection. Engagement is specifically assessed with the number of days over which the app was opened by participants.
Engagement with program - number of weeks with app openings | 6 months (26 weeks)
  Collected via back-end app data collection. Engagement is specifically assessed with the number of weeks over which the app was opened by participants.
Engagement with program - average duration of app sessions | 6 months (26 weeks)
  Collected via back-end app data collection. Engagement is specifically assessed with the average duration of app sessions completed by participants. Outcome unit of measure = duration in minutes.
Engagement with program - use of app features | 6 months (26 weeks)
  Collected via back-end app data collection. Engagement is specifically assessed with the use of app features (practice quits, challenges, logging vape sessions) by participants. Reported as the number of times each app feature was used.
Engagement with coach | 6 months (26 weeks)
  Collected via back-end app data collection. Engagement is specifically assessed with average number of messages sent by coach to participant per week and average number of messages sent by participant to coach per week.
Average number of weeks with coach engagement | 6 months (26 weeks)
  Collected via back-end app data collection. Specifically, the average number of weeks with at least one message sent from participant to coach.
Change in participant self-reported health | 6 months (26 weeks)
  Participant health is assessed with the following: "Would you say that in general your health is... Select one" And the following choices: "Excellent", "Very good", "Good", "Fair", and "Poor"
Use of other vaping cessation tools | 6 months (26 weeks)
  Assessed via self-report. Participants are asked about other vaping cessation tools they have used throughout the last 6 months. Tools asked about include: apps (other than Pivot), counseling, medications, acupuncture, hypnotherapy, etc. Participants can report other tools not included in the list provided. Outcome reported as the number of participants who have used each other vaping cessation tool.
Alcohol use behavior | 12, 26, and 52 weeks
  Assessed via the Alcohol Use Disorders Identification Test-Concise (AUDIT-C) screening questionnaire, 3 items. A score is calculated from a sum of the 3 items. Possible scores on the scale range from 0-12. A score of 0 indicates no alcohol use. Higher scores indicate greater alcohol use behavior, a worse outcome.
Presence of depressive symptoms | 12, 26, and 52 weeks
  Assessed via the Center of Epidemiological Studies Depression Scale (CES-D) screening questionnaire, 10 items. A score is calculated from a sum of the 10 items. Possible scores on the scale range from 0-30. Higher scores indicate greater severity of depressive symptoms, a worse outcome.
Living environment relating to vaping and cigarette smoking | 12, 26, and 52 weeks
  Assessed via participant self-report of living with other adults who vape and/or smoke, living with a romantic partner who vapes and/or smokes. Participants asked: "Of the adults you live with, how many smoke cigarettes?" and "Of the adults you live with, how many vape/use e-cigs?". Outcome unit of measure = number of adults.
Living/relationship environment relating to vaping and cigarette smoking | 12, 26, and 52 weeks
  Assessed via participant self-report of living with a romantic partner who vapes and/or smokes. Participants asked: "Do you live with a romantic partner who smokes cigarettes?" (yes/no) and "Do you live with a romantic partner who vapes/uses e-cigs?" (yes/no). Outcomes measure reported as number of participants who live with a romantic partner that smokes, and number that live with a romantic partner that vapes (participants that answer yes to these questions).
Social environment relating to vaping and cigarette smoking | 12, 26, and 52 weeks
  Assessed via participant self-report of the number of their close friends who vape and/or smoke. Participants asked: "How many of your close friends smoke cigarettes?" and "How many of your close friends vape/use e-cigs?". Outcome unit of measure = number of close friends.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Marler, MD, Principal Investigator — Pivot Health Technologies Inc.
Locations (1):
- Pivot Health Technologies, Inc., San Carlos, California, United States

REFERENCES:
- [Derived] Marler JD, Fujii CA, Utley MT, Balbierz DJ, Galanko JA, Utley DS. Outcomes of a Comprehensive Mobile Vaping Cessation Program in Adults Who Vape Daily: Cohort Study. JMIR Form Res. 2024 Oct 28;8:e57376. doi: 10.2196/57376. PMID 39331522